CLINICAL TRIAL: NCT02831855
Title: A PHASE 3B/4 RANDOMIZED DOUBLE BLIND PLACEBO CONTROLLED STUDY OF METHOTREXATE (MTX) WITHDRAWAL IN SUBJECTS WITH RHEUMATOID ARTHRITIS (RA) TREATED WITH TOFACITINIB 11MG MODIFIED RELEASE (MR) FORMULATION
Brief Title: Methotrexate Withdrawal Study of Tofacitinib Modified Release Formulation in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921192; 2016-001825-15 (EudraCT Number)
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Tofacitinib; CP-690,550; Xeljanz; methotrexate withdrawal; withdrawal study
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CP-690,550 and methotrexate (Experimental): Open-label tofacitinib tablet and blinded methotrexate capsule
  Interventions: Drug: CP-690,550; Drug: Methotrexate
- CP-690,550 and placebo (Placebo Comparator): open-label tofacitinib tablet and blinded matching placebo for methotrexate capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP-690,550 — During the open-label run-in phase (Day 1 to Week 24), all subjects will receive one tablet open-label tofacitinib MR 11mg orally QD and open-label methotrexate capsule(s) orally every week at prior stabilized dose.
  During the double-blind phase, subjects who are randomized to the treatment arm will receive the same dosage of tofacitinib and methotrexate as describe above.
  Other Names: tofacitinib
  Arms: CP-690,550 and methotrexate
Drug: Methotrexate — During the open-label run-in phase (Day 1 to Week 24), all subjects will receive one tablet open-label tofacitinib MR 11mg orally QD and open-label methotrexate capsule(s) orally every week at prior stabilized dose.
  During the double-blind phase, subjects who are randomized to the treatment arm will receive the same dosage of tofacitinib and methotrexate as describe above.
  Arms: CP-690,550 and methotrexate
Drug: Placebo — During the double-blind phase, subjects who are randomized to the comparison arm will receive 11mg QD tofacitinib and the placebo capsules matching for methotrexate.
  Arms: CP-690,550 and placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of tofacitinib modified release formulation (11mg QD) versus tofacitinib modified release formulation plus continued methotrexate treatment in subjects with moderate to severe rheumatoid arthritis who are insufficiently responding to their stable dose of methotrexate treatment.

ELIGIBILITY:
Key Inclusion Criteria

- Must be 18 years of age or older.

Have a score of 6 or greater on the 2010 American College of Rheumatology/European League Against Rheumatism Classification Criteria for Rheumatoid Arthritis at and/or prior to Screening Visit.

* Have ≥4 tender/painful joints on motion and ≥4 swollen joints (28 joint counts) at both Screening Visit and Baseline Visit (Visit 1).
* Have moderate to severe disease activity as defined by CDAI>10 and DAS28-4(ESR) ≥3.2 at Baseline Visit.
* Have taken an oral MTX treatment regimen (15-25mg/week) continuously for at least 4 months prior to the screening visit and has taken a stable weekly dose of oral MTX with supplemental folic acid or folinic acid for at least 4 weeks prior to the baseline visit (conversion from parenteral MTX to oral MTX will require stabilization of the treatment regimen for at least 1 month).
* Subjects must screen negative for active tuberculosis or inadequately treated tuberculosis infection (active or latent).

Key Exclusion Criteria

* Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children and female subjects of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 3 months after the last dose of investigational product.
* Subjects with infection or infection history; subjects with any current malignancy or a history of malignancy (except adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ); subjects with history of, or current evidence for, severe gastrointestinal narrowing (pathologic or iatrogenic); and subjects with history of documented diverticulitis.
* Subjects with a history of insufficient response to ≥2 biologics, regardless of the class.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (135):
- United States (59):
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Arthrocare, Arthritiscare & Research, PC, Gilbert, Arizona
  - SunValley Arthritis Center, Ltd., Peoria, Arizona
  - CHI St. Vincent Medical Group Hot Springs, Hot Springs, Arkansas
  - Med Investigations, Inc, Fair Oaks, California
  - HCP Clinical Research, LLC, Huntington Beach, California
  - Sierra Rheumatology, Roseville, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Robin K. Dore, MD, Inc., Tustin, California
  - Inland Rheumatology and Osteoporosis Medical Group, Upland, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Desert Valley Medical Group, Victorville, California
  - AARDS Research Inc, Aventura, Florida
  - RASF-Clinical Research Inc, Boca Raton, Florida
  - Omega Research Consultants, DeBary, Florida
  - University of Florida College of Medicine - Jacksonville - Rheumatology Research, Jacksonville, Florida
  - University of Florida, Rheumatology at ACC, Jacksonville, Florida
  - Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - Jeffrey Alper, MD, Naples, Florida
  - Medallion Clinical Research Institute, LLC, Naples, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Florida Arthritis & Osteoporosis Center, Port Richey, Florida
  - Gulf Coast Medical Center, Port Richey, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - USF Health Morsani Center for Advanced Healthcare, Tampa, Florida
  - BayCare Medical Group, Inc, Tampa, Florida
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Quincy Medical Group, Quincy, Illinois
  - Beacon Medical Group Rheumatology Main Street, Granger, Indiana
  - Diagnostic Rheumatology and Research, PC, Indianapolis, Indiana
  - Ochsner Clinic Baton Rouge, Baton Rouge, Louisiana
  - Phase III Clinical Research, Fall River, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Bronson Internal Medicine and Rheumatology, Battle Creek, Michigan
  - Western Michigan University Homer Stryker MD, Kalamazoo, Michigan
  - North Mississippi Medical Clinics, Inc. - Clinical Research, Tupelo, Mississippi
  - Arthritis & Osteoporosis Associates, Freehold, New Jersey
  - Radnet, Marlton, New Jersey
  - Arthritis, Rheumatic & Back Disease Associates, P.A., Voorhees Township, New Jersey
  - Open MRI & Diagnostic Imaging of Wall, Wall, New Jersey
  - AAIR Research Center, Rochester, New York
  - Physicians East, PA, Greenville, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Trinity Health Center-Medical Arts, Minot, North Dakota
  - Group Health Associates, Cincinnati, Ohio
  - Cincinnati Rheumatic Disease Study Group, Inc., Cincinnati, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation (OMRF), Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, P.C., Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Piedmont Arthritis Clinic, Greenville, South Carolina
  - Articularis Healthcare Group dba ACME Research, Orangeburg, South Carolina
  - Articularis Healthcare Group d/b/a Low Country Rheumatology, Summerville, South Carolina
  - Pioneer Research Solutions, Inc., Cypress, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Center for Arthritis and Rheumatic Diseases, Chesapeake, Virginia
  - Center for Arthritis and Rheumatic Diseases, Suffolk, Virginia
- Australia (4):
  - Genesis Research Services Pty Ltd, Broadmeadow, New South Wales
  - Optimus Clinical Research Pty Ltd, Kogarah, New South Wales
  - Rheumatology Research Unit, Maroochydore, Queensland
  - Emeritus Research, Melbourne, Victoria
- Belgium (2):
  - ReumaClinic, Genk
  - AZ Delta, Roeselare
- Bulgaria (6):
  - University Multiprofile Hospital for Active Treatment Dr. G. Stranski EAD, Pleven
  - Multiprofile Hospital for Active Treatment - Plovdiv AD, Rheumatology Department, Plovdiv
  - Multiprofile Hospital for Active Treatment Trimontium OOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment - Kaspela EOOD, Plovdiv
  - National Multiprofile Transport Hospital Tsar Boris III, Sofia
  - Medical Centre Synexus Sofia EOOD, Sofia
- Czechia (12):
  - CCBR Czech Brno, s.r.o., Brno, Czech Republic
  - LEKARNA LANCIER s.r.o., Brno
  - Lekarna Na Lidicke, Brno
  - Revmacentrum MUDr. Mostera, s.r.o., Revmatologie a interna, Brno
  - CCBR Ostrava, s.r.o., Ostrava
  - Lekarna Rezidence Nova Karolina, Ostrava
  - Revmatologicky ustav, Lekrna, Prague
  - Revmatologicky ustav, Prague
  - Lekarna Hradebni s.r.o., Uherské Hradiště
  - MEDICAL PLUS, s.r.o. Revmatologicka a osteologicka ambulance, Uherské Hradiště
  - PV - MEDICAL s.r.o., Revmatologicka ambulance, Zlín
  - Revmavita s.r.o, Lekarna, Zlín
- Hamburger Rheuma Forschungszentrum I, Hamburg, Germany
- Hungary (4):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Revita Rendelo, Budapest
  - Qualiclinic Kft., Budapest
  - CRU Hungary Kft., Miskolc
- Mexico (2):
  - Morales Vargas Centro de Investigacion SC (Consultorio Anexo), León, Guanajuato
  - Centro de Investigacion y Tratamiento Reumatologico SC Consultorio Medico de Reumatologia (CINTRE), Mexico City, Mexico City
- Philippines (2):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - Far Eastern University - Nicanor Reyes Medical Foundation, Marian Medical Arts Bldg, Quezon City, National Capital Region
- Poland (7):
  - Zdrowie OSTEO-MEDIC s.c. L i A. Racewicz, A i J. Supronik, Bialystok
  - ClinicMed Daniluk, Nowak. Sp. j., Bialystok
  - Nzoz Bif - Med, Bytom
  - Centrum Medyczne Pratia Krakow, Krakow
  - Malopolskie Centrum Medyczne S.C., Krakow
  - NZOZ Lecznica MAK-MED. S.C., Nadarzyn
  - MTZ Clinical Research Sp. z o.o., Warsaw
- Russia (8):
  - Federal State Budgetary Scientific Institution "Research Institute of Rheumatology, Moscow
  - FSBEI HE "Orenburg State Medical University" of MoH RF, Orenburg
  - FSBIH "Clinical Hospital #122 n.a. L.G. Sokolov" of FMBA of Russia, Saint Petersburg
  - SPb SBIH "Consultative-Diagnostic Centre #85", Saint Petersburg
  - SBIH "Samara Regional Clinical Hospital n.a. V.D. Seredavin", Samara
  - NSHI "Departmental Hospital at Smolensk station OJSC "Russian Railways", Smolensk
  - SAHI YR Clinical Hospital of Emergency Medical Care n.a. N.V. Soloviev, Yaroslavl
  - State Budgetary Institution of Healthcare of Yaroslavl Region "Regional Clinical Hospital", Yaroslavl
- Slovakia (5):
  - AAGS s.r.o., Dunajská Streda
  - MEDMAN s.r.o., Martin
  - REUMACENTRUM s.r.o., Partizánske
  - MUDr. Zuzana Cizmarikova, s.r.o., Poprad
  - Reumex s.r.o, Rimavská Sobota
- St. Augustine's Hospital, Durban, KwaZulu-Natal, South Africa
- South Korea (7):
  - Clinical Trial Pharmacy, KyungHee University Hospital, Seoul
  - KyungHee University Hospital, Seoul
  - CTC Pharmacy, Seoul National University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Clinical Trial Pharmacy, The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea Seoul, St. Mary's Hospital, Seoul
- Spain (3):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruna
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital Infanta Luisa, Seville
- United Kingdom (12):
  - Countess of Chester Hospital NHS Foundation Trust, Chester, Cheshire
  - Pharmacy (dispensary), Chester, Cheshire
  - Countess of Chester Hospital NHS Foundation Trust, Ellesmere Port, Cheshire
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire
  - Pharmacy, Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire
  - Department of Rheumatology, Wirral University Teaching Hospital NHS Foundation Trust, Metropolitan Borough of Wirral, Merseyside
  - Pharmacy Department, Wirral University Teaching Hospital NHS Foundation Trust, Metropolitan Borough of Wirral, Merseyside
  - Wirral University Teaching Hospital NHS Foundation Trust, Metropolitan Borough of Wirral, Merseyside
  - Pharmacy Department, Dudley, WEST Midlands
  - The Dudley Group NHS Foundation Trust, Dudley, WEST Midlands
  - Pharmacy, Manchester
  - University Hospital of South Manchester NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Background] Karaman MW, Herrgard S, Treiber DK, Gallant P, Atteridge CE, Campbell BT, Chan KW, Ciceri P, Davis MI, Edeen PT, Faraoni R, Floyd M, Hunt JP, Lockhart DJ, Milanov ZV, Morrison MJ, Pallares G, Patel HK, Pritchard S, Wodicka LM, Zarrinkar PP. A quantitative analysis of kinase inhibitor selectivity. Nat Biotechnol. 2008 Jan;26(1):127-32. doi: 10.1038/nbt1358. PMID 18183025
- [Background] Meyer DM, Jesson MI, Li X, Elrick MM, Funckes-Shippy CL, Warner JD, Gross CJ, Dowty ME, Ramaiah SK, Hirsch JL, Saabye MJ, Barks JL, Kishore N, Morris DL. Anti-inflammatory activity and neutrophil reductions mediated by the JAK1/JAK3 inhibitor, CP-690,550, in rat adjuvant-induced arthritis. J Inflamm (Lond). 2010 Aug 11;7:41. doi: 10.1186/1476-9255-7-41. PMID 20701804
- [Background] Murray PJ. The JAK-STAT signaling pathway: input and output integration. J Immunol. 2007 Mar 1;178(5):2623-9. doi: 10.4049/jimmunol.178.5.2623. PMID 17312100
- [Background] O'Sullivan LA, Liongue C, Lewis RS, Stephenson SE, Ward AC. Cytokine receptor signaling through the Jak-Stat-Socs pathway in disease. Mol Immunol. 2007 Apr;44(10):2497-506. doi: 10.1016/j.molimm.2006.11.025. Epub 2007 Jan 17. PMID 17208301
- [Background] Fleischmann R, Cutolo M, Genovese MC, Lee EB, Kanik KS, Sadis S, Connell CA, Gruben D, Krishnaswami S, Wallenstein G, Wilkinson BE, Zwillich SH. Phase IIb dose-ranging study of the oral JAK inhibitor tofacitinib (CP-690,550) or adalimumab monotherapy versus placebo in patients with active rheumatoid arthritis with an inadequate response to disease-modifying antirheumatic drugs. Arthritis Rheum. 2012 Mar;64(3):617-29. doi: 10.1002/art.33383. PMID 21952978
- [Background] Fleischmann R, Kremer J, Cush J, Schulze-Koops H, Connell CA, Bradley JD, Gruben D, Wallenstein GV, Zwillich SH, Kanik KS; ORAL Solo Investigators. Placebo-controlled trial of tofacitinib monotherapy in rheumatoid arthritis. N Engl J Med. 2012 Aug 9;367(6):495-507. doi: 10.1056/NEJMoa1109071. PMID 22873530
- [Background] Kremer JM, Cohen S, Wilkinson BE, Connell CA, French JL, Gomez-Reino J, Gruben D, Kanik KS, Krishnaswami S, Pascual-Ramos V, Wallenstein G, Zwillich SH. A phase IIb dose-ranging study of the oral JAK inhibitor tofacitinib (CP-690,550) versus placebo in combination with background methotrexate in patients with active rheumatoid arthritis and an inadequate response to methotrexate alone. Arthritis Rheum. 2012 Apr;64(4):970-81. doi: 10.1002/art.33419. Epub 2011 Oct 17. PMID 22006202
- [Background] Kremer J, Li ZG, Hall S, Fleischmann R, Genovese M, Martin-Mola E, Isaacs JD, Gruben D, Wallenstein G, Krishnaswami S, Zwillich SH, Koncz T, Riese R, Bradley J. Tofacitinib in combination with nonbiologic disease-modifying antirheumatic drugs in patients with active rheumatoid arthritis: a randomized trial. Ann Intern Med. 2013 Aug 20;159(4):253-61. doi: 10.7326/0003-4819-159-4-201308200-00006. PMID 24026258
- [Background] Burmester GR, Benda B, Gruben D, Bradley J, Mebus C. Tofacitinib for rheumatoid arthritis - Authors' reply. Lancet. 2013 May 25;381(9880):1812-3. doi: 10.1016/S0140-6736(13)61115-0. No abstract available. PMID 23706795
- [Background] van Vollenhoven RF, Fleischmann R, Cohen S, Lee EB, Garcia Meijide JA, Wagner S, Forejtova S, Zwillich SH, Gruben D, Koncz T, Wallenstein GV, Krishnaswami S, Bradley JD, Wilkinson B; ORAL Standard Investigators. Tofacitinib or adalimumab versus placebo in rheumatoid arthritis. N Engl J Med. 2012 Aug 9;367(6):508-19. doi: 10.1056/NEJMoa1112072. PMID 22873531
- [Background] Felson DT, Smolen JS, Wells G, Zhang B, van Tuyl LH, Funovits J, Aletaha D, Allaart CF, Bathon J, Bombardieri S, Brooks P, Brown A, Matucci-Cerinic M, Choi H, Combe B, de Wit M, Dougados M, Emery P, Furst D, Gomez-Reino J, Hawker G, Keystone E, Khanna D, Kirwan J, Kvien TK, Landewe R, Listing J, Michaud K, Martin-Mola E, Montie P, Pincus T, Richards P, Siegel JN, Simon LS, Sokka T, Strand V, Tugwell P, Tyndall A, van der Heijde D, Verstappen S, White B, Wolfe F, Zink A, Boers M; American College of Rheumatology; European League Against Rheumatism. American College of Rheumatology/European League Against Rheumatism provisional definition of remission in rheumatoid arthritis for clinical trials. Arthritis Rheum. 2011 Mar;63(3):573-86. doi: 10.1002/art.30129. PMID 21294106
- [Background] Fries JF, Spitz PW, Young DY. The dimensions of health outcomes: the health assessment questionnaire, disability and pain scales. J Rheumatol. 1982 Sep-Oct;9(5):789-93. No abstract available. PMID 7175852
- [Background] Ware JE KM, Dewey JE. . How to score Version 2 of the SF 36 Health Survey (Standard & Acute forms). In: How to score Version 2 of the SF 36 Health Survey (Standard & Acute forms). Lincoln, Rhode Island: QualityMetric, Incorporated. 2000.
- [Background] Hurst NP, Kind P, Ruta D, Hunter M, Stubbings A. Measuring health-related quality of life in rheumatoid arthritis: validity, responsiveness and reliability of EuroQol (EQ-5D). Br J Rheumatol. 1997 May;36(5):551-9. doi: 10.1093/rheumatology/36.5.551. PMID 9189057
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Cella D, Lai JS, Chang CH, Peterman A, Slavin M. Fatigue in cancer patients compared with fatigue in the general United States population. Cancer. 2002 Jan 15;94(2):528-38. doi: 10.1002/cncr.10245. PMID 11900238
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Cohen SB, Pope J, Haraoui B, Irazoque-Palazuelos F, Korkosz M, Diehl A, Rivas JL, Lukic T, Liu S, Stockert L, Iikuni N, Keystone EC. Methotrexate withdrawal in patients with rheumatoid arthritis who achieve low disease activity with tofacitinib modified-release 11 mg once daily plus methotrexate (ORAL Shift): a randomised, phase 3b/4, non-inferiority trial. Lancet Rheumatol. 2019 Sep;1(1):e23-e34. doi: 10.1016/S2665-9913(19)30005-0. Epub 2019 Aug 6. PMID 38229356
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Fleischmann R, Haraoui B, Buch MH, Gold D, Sawyerr G, Shi H, Diehl A, Lee K. Analysis of Disease Activity Metrics in a Methotrexate Withdrawal Study among Patients with Rheumatoid Arthritis Treated with Tofacitinib plus Methotrexate. Rheumatol Ther. 2023 Apr;10(2):375-386. doi: 10.1007/s40744-022-00511-3. Epub 2022 Dec 19. PMID 36534208
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Cohen SB, Haraoui B, Curtis JR, Smith TW, Woolcott J, Gruben D, Murray CW. Impact of Methotrexate Discontinuation, Interruption, or Persistence in US Patients with Rheumatoid Arthritis Initiating Tofacitinib + Oral Methotrexate Combination. Clin Ther. 2022 Jul;44(7):982-997.e2. doi: 10.1016/j.clinthera.2022.05.002. Epub 2022 Jun 4. PMID 35667900
- [Derived] Cohen SB, Pope J, Haraoui B, Mysler E, Diehl A, Lukic T, Liu S, Stockert L, Germino R, Menon S, Shi H, Keystone EC. Efficacy and safety of tofacitinib modified-release 11 mg once daily plus methotrexate in adult patients with rheumatoid arthritis: 24-week open-label phase results from a phase 3b/4 methotrexate withdrawal non-inferiority study (ORAL Shift). RMD Open. 2021 Jun;7(2):e001673. doi: 10.1136/rmdopen-2021-001673. PMID 34103405
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921192

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label: Tofacitinib 11 mg + Methotrexate: Participants with moderate to severe rheumatoid arthritis (RA) and who were insufficiently responding to their stable dose of methotrexate treatment previous to enrollment in this study, received Tofacitinib modified release (MR) 11 milligram (mg) tablet once daily (QD) with methotrexate at their previous stable dose for 24 weeks in open label phase (OL).
- Double Blind: Tofacitinib 11 mg + Methotrexate Placebo: Participants with low disease activity (LDA) at the end of open label phase were randomized to receive Tofacitinib MR 11 mg tablet once daily with matching placebo to blinded methotrexate at their previously stabilized dose for 24 weeks in double blind phase.
- Double Blind: Tofacitinib 11mg + Methotrexate: Participants with LDA at the end of open label phase were randomized to receive Tofacitinib MR 11 mg tablet once daily with blinded methotrexate at their previously stabilized dose for 24 weeks in double blind phase.
Period: Open Label Phase (24 Weeks)
Arm/Group | Open Label: Tofacitinib 11 mg + Methotrexate | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Started | 694 | 0 | 0
Completed | 623 | 0 | 0
Not Completed | 71 | 0 | 0
Not completed — Adverse Event | 39 | 0 | 0
Not completed — Lost to Follow-up | 8 | 0 | 0
Not completed — Insufficient Clinical Response | 7 | 0 | 0
Not completed — Medication error,no linked adverse event | 2 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Not completed — Other | 4 | 0 | 0
Period: Double Blind Phase (24 Weeks)
Arm/Group | Open Label: Tofacitinib 11 mg + Methotrexate | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Started | 0 | 267 (Only eligible participants from open label phase, were randomized into double blind phase.) | 266 (Only eligible participants from open label phase, were randomized into double blind phase. .)
Treated | 0 | 264 | 266
Completed | 0 | 238 | 247
Not Completed | 0 | 29 | 19
Not completed — Adverse Event | 0 | 6 | 6
Not completed — Death | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Screen Failure | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 2
Not completed — Other | 0 | 2 | 5
Not completed — Insufficient Clinical Response | 0 | 6 | 1
Not completed — Protocol Violation | 0 | 5 | 2
Not completed — Randomized but not Treated | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Open-label phase safety analysis set (Safety-OL) included all participants who received at least 1 dose of Tofacitinib MR 11 mg plus Methotrexate during open-label phase.
Arm/Group | Open Label: Tofacitinib 11 mg + Methotrexate
Number analyzed (Participants) | 694
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.77 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 532
  Male | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59
  Not Hispanic or Latino | 635
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 37
  Black or African American | 33
  White | 594
  Others | 30

OUTCOME MEASURES:

1. Primary Outcome: Double Blind Phase: Change From Randomization in Disease Activity Score in 28 Joints Using 4 Variables (DAS28-4) (Erythrocyte Sedimentation Rate [ESR]) at Week 48
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from swollen joint count (SJC) and tender/painful joint count (TJC) using 28 joints count, ESR (millimeters per hour [mm/hr]) and participant global assessment of arthritis (PtGA) on a 100 millimeter (mm) visual analog scale (VAS: scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicate worse health condition). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (ESR) less than or equal to (<=) 3.2 implied low disease activity and greater than (>) 3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (ESR) less than (<) 2.6 implied remission. DAS28-4 (ESR) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*In(ESR in mm/hour) + 0.014*PtGA in mm; ln = natural logarithm, sqrt = square root of.
Time Frame: Randomization (last non-missing measurement on or prior to the first dosing date in DB phase at Week 24), Week 48
Population: Double-Blind Period Full Analysis Set (FAS-DB) included all participants who received at least 1 dose of investigational drug during the OL phase, were randomized and received at least 1 dose of the randomized investigational drug regimen during DB phase. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 235 | 237
units on a scale | 0.33 (0.07) | 0.03 (0.07)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Linear mixed-effect model of repeated measures (MMRM) was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a biological disease-modifying anti-rheumatic drug (bDMARD), and baseline DAS28-4 (ESR) value as a covariate; Test type: Non-Inferiority — Non-inferiority (NI) of Tofacitinib 11 mg + Methotrexate Placebo to Tofacitinib 11 mg + continued Methotrexate was concluded if the upper bound of 95% 2-sided confidence interval (CI) for difference between the 2 arms (Tofacitinib 11 mg + Methotrexate Placebo reporting arm - Tofacitinib 11 mg + continued Methotrexate arm) was lower than 0.6; p = 0.0005, MMRM — The p-value is one-sided for the test against the NI margin of 0.6; Least Square (LS) Mean Difference = 0.30, 95% CI 2-sided [0.12 to 0.48], Standard Error of Mean 0.09

2. Secondary Outcome: Double Blind Phase: Change From Randomization in DAS28-4 ESR at Week 36
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hr) and PtGA on a 100 millimeter (mm) VAS (VAS: scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicate worse health condition). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (ESR) less than or equal to (<=) 3.2 implied low disease activity and greater than (>) 3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (ESR) less than (<) 2.6 implied remission. DAS28-4 (ESR) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*In(ESR in mm/hour) + 0.014*PtGA in mm; ln = natural logarithm, sqrt = square root of.
Time Frame: Randomization (last non-missing measurement on or prior to the first dosing date in DB phase at Week 24), Week 36
Population: FAS-DB included all participants who received at least 1 dose of investigational drug during the OL phase, were randomized and received at least 1 dose of the randomized investigational drug regimen during DB phase. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 253 | 253
units on a scale | 0.40 (0.07) | 0.18 (0.07)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD and baseline DAS28-4 (ESR) value as a covariate; Test type: Superiority; LS Mean Difference = 0.22, 95% CI 2-sided [0.03 to 0.41], Standard Error of Mean 0.10

3. Secondary Outcome: Double Blind Phase: Change From Randomization in DAS28-4 (C-reactive Protein [CRP]) at Weeks 36 and 48
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated from SJC and TJC using 28 joints count, CRP (milligrams per liter [mg/L]) and PtGA on a 100 mm VAS (VAS: scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicate worse health condition). Total DAS28-4 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (CRP) <= 3.2 implied low disease activity and > 3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (CRP) < 2.6 implied remission. DAS28-4 (CRP) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP in mg/L +1) + 0.014*PtGA in mm+ 0.96; ln = natural logarithm, sqrt = square root of.
Time Frame: Randomization (last non-missing measurement on or prior to the first dosing date in DB phase at Week 24), Weeks 36 and 48
Population: FAS-DB was analyzed. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
units on a scale
  Change at Week 36: number analyzed (Participants) | 250 | 254
  Change at Week 36 | 0.38 (0.06) | 0.13 (0.06)
  Change at Week 48: number analyzed (Participants) | 231 | 235
  Change at Week 48 | 0.29 (0.06) | 0.01 (0.06)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Linear MMRM was used that included the fixed effects of treatment, visit, treatment -by-visit interaction, prior use of a bDMARD and baseline DAS28-4 (CRP) value as a covariate; Test type: Superiority; LS Mean Difference = 0.26, 95% CI 2-sided [0.08 to 0.43], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Linear MMRM was used that included the fixed effects of treatment, visit, treatment -by-visit interaction, prior use of a bDMARD and baseline DAS28-4 (CRP) value as a covariate; Test type: Superiority; LS Mean Difference = 0.28, 95% CI 2-sided [0.11 to 0.45], Standard Error of Mean 0.09

4. Secondary Outcome: Double Blind Phase: Change From Randomization in Clinical Disease Activity Index (CDAI) at Weeks 36 and 48
Description: CDAI was calculated from tender and swollen joints using 28 joint count, PtGA and physician global assessment of arthritis (PhyGA). PtGA and PhyGA both were assessed on 0-10 centimeter (cm) VAS scale (VAS: scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). CDAI total score ranged from 0 to 76, where higher scores indicated higher disease activity. CDAI score of <=10 indicated low disease activity and a score of <= 2.8 indicated remission. CDAI = (28TJC) + (28SJC) + (PhyGA in cm) + (PtGA in cm).
Time Frame: as for outcome 3
Population: FAS-DB was analyzed. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
units on a scale
  Change at Week 36: number analyzed (Participants) | 254 | 259
  Change at Week 36 | 3.58 (0.49) | 1.84 (0.48)
  Change at Week 48: number analyzed (Participants) | 238 | 244
  Change at Week 48 | 2.97 (0.48) | 0.84 (0.47)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD and baseline CDAI value as a covariate; Test type: Superiority; LS Mean Difference = 1.74, 95% CI 2-sided [0.40 to 3.07], Standard Error of Mean 0.68
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD and baseline CDAI value as a covariate; Test type: Superiority; LS Mean Difference = 2.13, 95% CI 2-sided [0.83 to 3.43], Standard Error of Mean 0.66

5. Secondary Outcome: Double Blind Phase: Change From Randomization in Simplified Disease Activity Index (SDAI) at Weeks 36 and 48
Description: SDAI was calculated from tender and swollen joints using 28 joint count, PtGA, PhyGA and CRP (in mg/dL). PtGA and PhyGA both were assessed on 0-10 cm VAS scale (VAS: scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). SDAI total score ranged from 0 to 86, where higher scores indicated higher disease activity. SDAI score of <=11 indicates low disease activity and a score of <=3.3 indicates remission. SDAI = (28TJC) + (28SJC) + (PhyGA in cm) + (PtGA in cm) + (CRP in mg/dL).
Time Frame: as for outcome 3
Population: FAS-DB was analyzed. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
units on a scale
  Change at Week 36: number analyzed (Participants) | 249 | 254
  Change at Week 36 | 3.83 (0.52) | 1.88 (0.51)
  Change at Week 48: number analyzed (Participants) | 231 | 235
  Change at Week 48 | 3.16 (0.50) | 0.94 (0.49)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD and baseline SDAI value as a covariate; Test type: Superiority; LS Mean Difference = 1.95, 95% CI 2-sided [0.53 to 3.37], Standard Error of Mean 0.72
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD and baseline SDAI value as a covariate; Test type: Superiority; LS Mean Difference = 2.23, 95% CI 2-sided [0.86 to 3.59], Standard Error of Mean 0.69

6. Secondary Outcome: Double Blind Phase: Percentage of Participants With Low Disease Activity (LDA) Assessed by DAS28-4 (ESR) Less Than or Equal to (<=) 3.2 at Weeks 36 and 48
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hr) and PtGA on a 100 mm VAS (VAS: scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicated worse health condition). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (ESR) <=3.2 implied low disease activity and >3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (ESR) <2.6 implied remission. DAS28-4 (ESR) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*In(ESR in mm/hour) + 0.014*PtGA in mm; ln = natural logarithm, sqrt = square root of.
Time Frame: Weeks 36 and 48
Population: FAS-DB included all participants who received at least 1 dose of investigational drug during the OL phase, were randomized and received at least 1 dose of the randomized investigational drug regimen during DB phase. Non-responder imputation (NRI) method was used to impute missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 42.42 | 48.12
  Week 48 | 45.08 | 49.62
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -5.69, 95% CI 2-sided [-14.15 to 2.76]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -4.54, 95% CI 2-sided [-13.04 to 3.94]

7. Secondary Outcome: Double Blind Phase: Percentage of Participants With LDA Assessed by DAS28-4 (CRP) <=3.2 at Weeks 36 and 48
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated from SJC and TJC using 28 joints count, CRP (mg/L) and PtGA on a 100 mm VAS (VAS: scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicate worse health condition). Total DAS28-4 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (CRP) <=3.2 implied low disease activity and >3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (CRP) <2.6 implied remission. DAS28-4 (CRP) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP in mg/L +1) + 0.014*PtGA in mm+ 0.96; ln = natural logarithm, sqrt = square root of.
Time Frame: Weeks 36 and 48
Population: FAS-DB included all participants who received at least 1 dose of investigational drug during the OL phase, were randomized and received at least 1 dose of the randomized investigational drug regimen during DB phase. NRI method was used to impute missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 65.53 | 70.68
  Week 48 | 65.91 | 74.44
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -5.14, 95% CI 2-sided [-13.07 to 2.77]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -8.52, 95% CI 2-sided [-16.28 to -0.76]

8. Secondary Outcome: Double Blind Phase: Percentage of Participants With LDA Assessed by CDAI <=10 at Weeks 36 and 48
Description: CDAI was calculated from tender and swollen joints using 28 joint count, PtGA and PhyGA. PtGA and PhyGA both were assessed on 0-10 cm VAS scale (VAS: scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). CDAI total score ranged from 0 to 76, where higher scores indicated higher disease activity. CDAI score of <=10 indicated low disease activity and a score of <= 2.8 indicated remission. Percentage of participants with CDAI <=10 were reported. CDAI = (28TJC) + (28SJC) + (PhyGA in cm) + (PtGA in cm).
Time Frame: Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 66.29 | 73.68
  Week 48 | 65.15 | 77.07
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -7.39, 95% CI 2-sided [-15.17 to 0.38]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -11.91, 95% CI 2-sided [-19.56 to -4.26]

9. Secondary Outcome: Double Blind Phase: Percentage of Participants With LDA Assessed by SDAI <=11 at Weeks 36 and 48
Description: SDAI was calculated from tender and swollen joints using 28 joint count, PtGA, PhyGA and CRP (in mg/dL). PtGA and PhyGA both were assessed on 0-10 cm VAS scale (VAS: scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). SDAI total score ranged from 0 to 86, where higher scores indicated higher disease activity. SDAI score of <=11 indicated low disease activity and a score of <=3.3 indicated remission. SDAI = (28TJC) + (28SJC) + (PhyGA in cm) + (PtGA in cm) + (CRP in mg/dL).
Time Frame: Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 66.29 | 73.31
  Week 48 | 66.29 | 76.32
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -7.02, 95% CI 2-sided [-14.81 to 0.77]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -10.02, 95% CI 2-sided [-17.68 to -2.37]

10. Secondary Outcome: Double Blind Phase: Percentage of Participants With Remission Assessed by American College of Rheumatology-European League Against Rheumatism (ACR-EULAR) Boolean at Weeks 36 and 48
Description: ACR-EULAR Boolean remission was when a participant satisfied all of the following: tender joint count, swollen joint count (both based on a 28-joint assessment), CRP (in mg/dL), and PtGA (VAS: 0 cm [very well] to 10 cm [worst], higher scores indicated worse health condition) and all scores were <=1.
Time Frame: Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 15.53 | 24.06
  Week 48 | 22.35 | 23.68
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -8.52, 95% CI 2-sided [-15.27 to -1.78]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Two Sided; Difference in percentage of participants = -1.33, 95% CI 2-sided [-8.50 to 5.83]

11. Secondary Outcome: Double Blind Phase: Percentage of Participants With Remission Assessed by DAS28-4 (ESR) Less Than [<] 2.6 at Weeks 36 and 48
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hr) and PtGA on a 100 mm VAS (VAS: scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicate worse health condition). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity and >3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (ESR) <2.6 implied remission. DAS28-4 (ESR) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.70*In(ESR in mm/hour) + 0.014*PtGA in mm. Percentage of participants with DAS remission (DAS28-4-ESR<2.6) were reported in this outcome measure.
Time Frame: Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 20.45 | 28.57
  Week 48 | 23.86 | 30.08
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -8.11, 95% CI 2-sided [-15.40 to -0.82]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -6.21, 95% CI 2-sided [-13.74 to 1.32]

12. Secondary Outcome: Double Blind Phase: Percentage of Participants With Remission Assessed by DAS28-4 (CRP) <2.6 at Weeks 36 and 48
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated from SJC and TJC using 28 joints count, CRP (mg/L) and PtGA on a 100 mm VAS (VAS: scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicate worse health condition). Total DAS28-4 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (CRP) <=3.2 implied low disease activity and >3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (CRP) <2.6 implied remission. DAS28-4 (CRP) = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP in mg/l +1) + 0.014*PtGA in mm+ 0.96. Percentage of participants with DAS remission (DAS28-4-CRP<2.6) were reported in this outcome measure.
Time Frame: Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 50.00 | 55.64
  Week 48 | 50.38 | 54.51
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -5.63, 95% CI 2-sided [-14.12 to 2.84]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -4.13, 95% CI 2-sided [-12.62 to 4.36]

13. Secondary Outcome: Double Blind Phase: Percentage of Participants With Remission Assessed by CDAI <=2.8 at Weeks 36 and 48
Description: CDAI was calculated from tender and swollen joints using 28 joint count, PtGA and PhyGA. PtGA and PhyGA both were assessed on 0-10 cm VAS scale (VAS: scores ranging from 0 cm [very well] to 10 cm [worst]), where higher scores indicated greater affliction due to disease activity). CDAI total score ranged from 0 to 76, where higher scores indicated higher disease activity. CDAI score of <=10 indicated low disease activity and a score of <= 2.8 indicated remission. CDAI = (28TJC) + (28SJC) + (PhyGA in cm) + (PtGA in cm).
Time Frame: Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 23.48 | 32.33
  Week 48 | 28.41 | 30.83
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -8.84, 95% CI 2-sided [-16.44 to -1.24]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -2.41, 95% CI 2-sided [-10.18 to 5.35]

14. Secondary Outcome: Double Blind Phase: Percentage of Participants With Remission Assessed by SDAI <=3.3 at Weeks 36 and 48
Description: as for outcome 5
Time Frame: Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 22.73 | 31.58
  Week 48 | 28.79 | 31.95
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -8.85, 95% CI 2-sided [-16.38 to -1.31]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -3.16, 95% CI 2-sided [-10.99 to 4.65]

15. Secondary Outcome: Double Blind Phase: Percentage of Participants Achieving an American College of Rheumatology 20 Percent (%) (ACR20) Response at Weeks 36 and 48
Description: Participants with 20% improvement in tender and swollen joint counts and 20% improvement in at least 3 of the 5 measures: PtGA, PhyGA, participant's assessment of arthritis pain, Health Assessment Questionnaire-Disability Index (HAQ-DI) and CRP. PtGA: participant assessed health on VAS, 0 mm (very well) to 100 mm (worst health condition), higher scores = worse condition. PhyGA: physician judged participants' pain on VAS, 0 (no pain) to 100 mm (extreme pain), higher scores = more pain. Participant's assessment of arthritis pain: participant assessed pain on VAS, 0 mm (no pain) to 100 mm (most severe pain), higher score = more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score implied more disability. The improvement was relative to baseline (Day 1).
Time Frame: Baseline (Day 1), Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 73.86 | 80.83
  Week 48 | 73.11 | 79.70
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -6.96, 95% CI 2-sided [-14.06 to 0.14]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -6.59, 95% CI 2-sided [-13.80 to 0.61]

16. Secondary Outcome: Double Blind Phase: Percentage of Participants Achieving an American College of Rheumatology 50% (ACR50) Response at Weeks 36 and 48
Description: Participants with 50% improvement in tender and swollen joint counts and 50% improvement in at least 3 of the 5 measures: PtGA, PhyGA, participant's assessment of arthritis pain, HAQ-DI and CRP. PtGA: participant assessed health on VAS, 0 mm (very well) to 100 mm (worst health condition), higher scores = worse condition. PhyGA: physician judged participants' pain on VAS, 0 (no pain) to 100 mm (extreme pain), higher scores = more pain. Participant's assessment of arthritis pain: participant assessed pain on VAS, 0 mm (no pain) to 100 mm (most severe pain), higher score = more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score implied more disability. The improvement was relative to baseline (Day 1).
Time Frame: Baseline (Day 1), Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 53.79 | 66.54
  Week 48 | 55.30 | 67.29
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -12.75, 95% CI 2-sided [-21.01 to -4.48]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -11.99, 95% CI 2-sided [-20.22 to -3.75]

17. Secondary Outcome: Double Blind Phase: Percentage of Participants Achieving an American College of Rheumatology 70% (ACR70) Response at Weeks 36 and 48
Description: Participants with 70% improvement in tender and swollen joint counts and 70% improvement in at least 3 of the 5 measures: PtGA, PhyGA, participant's assessment of arthritis pain, HAQ-DI and CRP. PtGA: participant assessed health on VAS, 0 mm (very well) to 100 mm (worst health condition), higher scores = worse condition. PhyGA: physician judged participants' pain on VAS, 0 (no pain) to 100 mm (extreme pain), higher scores = more pain. Participant's assessment of arthritis pain: participant assessed pain on VAS, 0 mm (no pain) to 100 mm (most severe pain), higher score = more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score implied more disability. The improvement was relative to baseline (Day 1).
Time Frame: Baseline (Day 1), Weeks 36 and 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 35.61 | 40.98
  Week 48 | 37.88 | 42.86
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -5.37, 95% CI 2-sided [-13.63 to 2.89]
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -4.97, 95% CI 2-sided [-13.32 to 3.36]

18. Secondary Outcome: Double Blind Phase: Change From Randomization in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Weeks 36 and 48
Description: HAQ-DI assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing/grooming; arising; eating; walking; reach; grip; hygiene; and other activities.. There were total of 30 items distributed in these 8 domains. Each item was scored on a 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 (least difficulty) and 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities.
Time Frame: as for outcome 3
Population: FAS-DB was analyzed. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
units on a scale
  Change at Week 36: number analyzed (Participants) | 252 | 259
  Change at Week 36 | 0.10 (0.03) | 0.01 (0.03)
  Change at Week 48: number analyzed (Participants) | 238 | 246
  Change at Week 48 | 0.01 (0.03) | 0.00 (0.03)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD and baseline HAQ-DI; Test type: Superiority; LS Mean Difference = 0.09, 95% CI 2-sided [0.02 to 0.16], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD and baseline HAQ-DI; Test type: Superiority; LS Mean Difference = 0.02, 95% CI 2-sided [-0.06 to 0.09], Standard Error of Mean 0.04

19. Secondary Outcome: Double Blind Phase: Change From Randomization in the Short Form 36 (SF-36) Health Survey 8 Domain Scores at Weeks 36 and 48
Description: SF-36 is a participant reported standardized survey designed to assess generic health related quality of life. It consisted of 36 items evaluating 8 aspects of functional health and well-being: physical functioning, role physical, bodily pain, social functioning, mental health, role emotional, vitality, and general health perception. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Scores of 8 health aspects were summarized to derive the 2 component scores (physical component scores [PCS], mental component scores [MCS]) ranging from 0 (worst) to 100 (best), where higher PCS/MCS indicated good health condition.
Time Frame: as for outcome 3
Population: FAS-DB was analyzed. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
units on a scale
  Change at Week 36: Physical Functioning: number analyzed (Participants) | 252 | 259
  Change at Week 36: Physical Functioning | -1.32 (0.50) | -0.88 (0.49)
  Change at Week 36: Role Physical Score: number analyzed (Participants) | 252 | 259
  Change at Week 36: Role Physical Score | -1.69 (0.48) | -0.02 (0.47)
  Change at Week 36: Social Functioning: number analyzed (Participants) | 252 | 259
  Change at Week 36: Social Functioning | -0.98 (0.50) | -0.84 (0.49)
  Change at Week 36: Bodily Pain Score: number analyzed (Participants) | 252 | 259
  Change at Week 36: Bodily Pain Score | -2.03 (0.53) | -0.58 (0.52)
  Change at Week 36: Mental Health Score: number analyzed (Participants) | 251 | 259
  Change at Week 36: Mental Health Score | -1.22 (0.51) | -0.32 (0.50)
  Change at Week 36: Role Emotional Score: number analyzed (Participants) | 252 | 259
  Change at Week 36: Role Emotional Score | -1.80 (0.56) | -0.69 (0.55)
  Change at Week 36: Vitality Score: number analyzed (Participants) | 251 | 259
  Change at Week 36: Vitality Score | -1.30 (0.50) | -0.15 (0.50)
  Change at Week 36: General Health Perception Score: number analyzed (Participants) | 252 | 259
  Change at Week 36: General Health Perception Score | -0.98 (0.44) | -0.87 (0.43)
  Change at Week 48: Physical Functioning: number analyzed (Participants) | 238 | 246
  Change at Week 48: Physical Functioning | -0.46 (0.49) | -0.97 (0.48)
  Change at Week 48: Role Physical Score: number analyzed (Participants) | 238 | 246
  Change at Week 48: Role Physical Score | -0.88 (0.51) | -0.15 (0.50)
  Change at Week 48: Social Functioning: number analyzed (Participants) | 238 | 246
  Change at Week 48: Social Functioning | -1.06 (0.53) | -0.55 (0.52)
  Change at Week 48: Bodily Pain Score: number analyzed (Participants) | 238 | 246
  Change at Week 48: Bodily Pain Score | -1.46 (0.54) | -0.71 (0.54)
  Change at Week 48: Mental Health Score: number analyzed (Participants) | 238 | 246
  Change at Week 48: Mental Health Score | -0.34 (0.54) | 0.12 (0.54)
  Change at Week 48: Role Emotional Score: number analyzed (Participants) | 238 | 246
  Change at Week 48: Role Emotional Score | -0.83 (0.54) | -0.36 (0.54)
  Change at Week 48: Vitality Score: number analyzed (Participants) | 238 | 246
  Change at Week 48: Vitality Score | -0.77 (0.52) | -0.25 (0.52)
  Change at Week 48: General Health Perception Score: number analyzed (Participants) | 238 | 246
  Change at Week 48: General Health Perception Score | -0.43 (0.45) | -1.05 (0.44)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Physical Functioning- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 physical component score as a covariate; Test type: Superiority; LS Mean Difference = -0.44, 95% CI 2-sided [-1.79 to 0.92], Standard Error of Mean 0.69
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Physical Functioning- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 physical component score as a covariate; Test type: Superiority; LS Mean Difference = 0.52, 95% CI 2-sided [-0.82 to 1.85], Standard Error of Mean 0.68
Statistical Analysis 3: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Role Physical Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 role physical score score as a covariate; Test type: Superiority; LS Mean Difference = -1.67, 95% CI 2-sided [-2.97 to -0.37], Standard Error of Mean 0.66
Statistical Analysis 4: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Role Physical Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 role physical score score as a covariate; Test type: Superiority; LS Mean Difference = -0.73, 95% CI 2-sided [-2.13 to 0.66], Standard Error of Mean 0.66
Statistical Analysis 5: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Social functioning- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 Social functioning score as a covariate; Test type: Superiority; LS Mean Difference = -0.14, 95% CI 2-sided [-1.50 to 1.21], Standard Error of Mean 0.69
Statistical Analysis 6: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Social functioning- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 Social functioning score as a covariate; Test type: Superiority; LS Mean Difference = -0.51, 95% CI 2-sided [-1.95 to 0.93], Standard Error of Mean 0.73
Statistical Analysis 7: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Bodily Pain Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 bodily pain score as a covariate; Test type: Superiority; LS Mean Difference = -1.45, 95% CI 2-sided [-2.90 to -0.01], Standard Error of Mean 0.74
Statistical Analysis 8: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Bodily Pain Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 bodily pain score as a covariate; Test type: Superiority; LS Mean Difference = -0.75, 95% CI 2-sided [-2.23 to 0.73], Standard Error of Mean 0.75
Statistical Analysis 9: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Mental Health Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 mental health score as a covariate; Test type: Superiority; LS Mean Difference = -0.90, 95% CI 2-sided [-2.29 to 0.49], Standard Error of Mean 0.71
Statistical Analysis 10: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Mental Health Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 mental health score as a covariate; Test type: Superiority; LS Mean Difference = -0.46, 95% CI 2-sided [-1.94 to 1.02], Standard Error of Mean 0.75
Statistical Analysis 11: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Role Emotional Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 role emotional score as a covariate; Test type: Superiority; LS Mean Difference = -1.11, 95% CI 2-sided [-2.64 to 0.43], Standard Error of Mean 0.78
Statistical Analysis 12: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Role Emotional Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 role emotional score as a covariate; Test type: Superiority; LS Mean Difference = -0.47, 95% CI 2-sided [-1.95 to 1.01], Standard Error of Mean 0.75
Statistical Analysis 13: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Vitality Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 vitality score as a covariate; Test type: Superiority; LS Mean Difference = -1.15, 95% CI 2-sided [-2.52 to 0.22], Standard Error of Mean 0.70
Statistical Analysis 14: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Vitality Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 vitality score as a covariate; Test type: Superiority; LS Mean Difference = -0.52, 95% CI 2-sided [-1.94 to 0.91], Standard Error of Mean 0.73
Statistical Analysis 15: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: General Health Perception Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 general health perception score as a covariate; Test type: Superiority; LS Mean Difference = -0.11, 95% CI 2-sided [-1.30 to 1.08], Standard Error of Mean 0.61
Statistical Analysis 16: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: General Health Perception Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 general health perception score as a covariate; Test type: Superiority; LS Mean Difference = 0.62, 95% CI 2-sided [-0.60 to 1.83], Standard Error of Mean 0.62

20. Secondary Outcome: Double Blind Phase: Change From Randomization in the SF-36 Health Survey Component Scores at Weeks 36 and 48
Description: SF-36 is a participant reported standardized survey designed to assess generic health related quality of life. It consisted of 36 items evaluating 8 aspects of functional health and well-being: physical functioning, role physical, bodily pain, social functioning, mental health, role emotional, vitality, and general health perception. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Scores of 8 health aspects were summarized aggregated to derive the two 2 component scores PCS and MCS ranging from 0 (worst) to 100 (best), where higher PCS/MCS indicated good health condition.
Time Frame: as for outcome 3
Population: FAS-DB was analyzed. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
units on a scale
  Change at Week 36: Physical Component Score: number analyzed (Participants) | 251 | 259
  Change at Week 36: Physical Component Score | -1.42 (0.44) | -0.60 (0.43)
  Change at Week 36: Mental Component Score: number analyzed (Participants) | 251 | 259
  Change at Week 36: Mental Component Score | -1.25 (0.48) | -0.43 (0.47)
  Change at Week 48: Physical Component Score: number analyzed (Participants) | 238 | 246
  Change at Week 48: Physical Component Score | -0.83 (0.44) | -0.92 (0.43)
  Change at Week 48: Mental Component Score: number analyzed (Participants) | 238 | 246
  Change at Week 48: Mental Component Score | -0.65 (0.51) | 0.03 (0.50)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Physical Component Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 physical component score- as a covariate; Test type: Superiority; LS Mean Difference = -0.82, 95% CI 2-sided [-2.01 to 0.37], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Physical Component Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a biological disease-modifying anti-rheumatic drug (DMARD), and baseline SF-36 physical component score- as a covariate; Test type: Superiority; LS Mean Difference = 0.09, 95% CI 2-sided [-1.11 to 1.29], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Mental Component Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 mental component score as a covariate; Test type: Superiority; LS Mean Difference = -0.82, 95% CI 2-sided [-2.13 to 0.49], Standard Error of Mean 0.67
Statistical Analysis 4: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Mental Component Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline SF-36 mental component score as a covariate; Test type: Superiority; LS Mean Difference = -0.68, 95% CI 2-sided [-2.06 to 0.70], Standard Error of Mean 0.70

21. Secondary Outcome: Double Blind Phase: Change From Randomization in the Work Productivity and Activity Impairment (WPAI) Scores at Week 36 and 48
Description: WPAI is 6-question participant rated questionnaire to determine the impact of rheumatoid arthritis and yields 4 types of outcomes: absenteeism (work time missed), presenteeism (impairment while working), work productivity loss (overall work impairment), and daily activity impairment (activity impairment) for a period of 7 days prior to a visit. These 4 outcomes are expressed as an impairment percentage (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Randomization (last non-missing measurement on or prior to the first dosing date in DB phase at Week 24), Week 36 and 48
Population: FAS-DB was analyzed. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time point.
Measure: Least Squares Mean (Standard Error); unit: percentage impairment
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage impairment
  Change at Week 36: Absenteeism: number analyzed (Participants) | 90 | 104
  Change at Week 36: Absenteeism | -1.39 (1.79) | -3.00 (1.69)
  Change at Week 36: Daily activity impairment: number analyzed (Participants) | 252 | 256
  Change at Week 36: Daily activity impairment | 4.00 (1.35) | 0.81 (1.34)
  Change at Week 36: Presenteeism: number analyzed (Participants) | 96 | 104
  Change at Week 36: Presenteeism | 3.68 (2.20) | 0.67 (2.07)
  Change at Week 36: Work productivity loss: number analyzed (Participants) | 90 | 101
  Change at Week 36: Work productivity loss | 3.03 (2.57) | 0.19 (2.41)
  Change at Week 48: Absenteeism: number analyzed (Participants) | 89 | 101
  Change at Week 48: Absenteeism | -2.21 (1.70) | -1.69 (1.61)
  Change at Week 48: Daily activity impairment: number analyzed (Participants) | 238 | 243
  Change at Week 48: Daily activity impairment | 2.86 (1.47) | 1.25 (1.46)
  Change at Week 48: Presenteeism: number analyzed (Participants) | 93 | 101
  Change at Week 48: Presenteeism | 2.82 (2.78) | 3.72 (2.61)
  Change at Week 48: Work productivity loss: number analyzed (Participants) | 89 | 98
  Change at Week 48: Work productivity loss | 2.98 (3.09) | 5.45 (2.91)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Absenteeism Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline WPAI absenteeism score as a covariate; Test type: Superiority; LS Mean Difference = 1.61, 95% CI 2-sided [-3.14 to 6.37], Standard Error of Mean 2.41
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Absenteeism Score- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline WPAI absenteeism score as a covariate; Test type: Superiority; LS Mean Difference = -0.51, 95% CI 2-sided [-5.01 to 3.99], Standard Error of Mean 2.28
Statistical Analysis 3: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Daily activity impairment- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline WPAI daily activity impairment score as a covariate; Test type: Superiority; LS Mean Difference = 3.19, 95% CI 2-sided [-0.51 to 6.89], Standard Error of Mean 1.88
Statistical Analysis 4: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Daily activity impairment- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline WPAI daily activity impairment score as a covariate; Test type: Superiority; LS Mean Difference = 1.60, 95% CI 2-sided [-2.41 to 5.61], Standard Error of Mean 2.04
Statistical Analysis 5: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Presenteeism- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline WPAI presenteeism score as a covariate; Test type: Superiority; LS Mean Difference = 3.01, 95% CI 2-sided [-2.84 to 8.87], Standard Error of Mean 2.97
Statistical Analysis 6: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Presenteeism- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline WPAI presenteeism score as a covariate; Test type: Superiority; LS Mean Difference = -0.90, 95% CI 2-sided [-8.34 to 6.54], Standard Error of Mean 3.77
Statistical Analysis 7: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Work productivity loss- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline WPAI work productivity loss score as a covariate; Test type: Superiority; LS Mean Difference = 2.84, 95% CI 2-sided [-3.97 to 9.65], Standard Error of Mean 3.45
Statistical Analysis 8: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Work productivity loss- Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline WPAI work productivity loss score as a covariate; Test type: Superiority; LS Mean Difference = -2.46, 95% CI 2-sided [-10.72 to 5.80], Standard Error of Mean 4.19

22. Secondary Outcome: Double Blind Phase: Change From Randomization in the European Quality of Life - 5 Dimensions Questionnaire (EQ-5D) Scores at Weeks 36 and 48
Description: EQ-5D was a participant completed instrument designed to assess impact on quality of life in terms of a single utility score in 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. 3 possible answers for mobility: 1=no problem in walking, 2=moderate problems in walking, 3= confined to bed; self-care: 1=no problem, 2=moderate problems, 3= unable to wash/dress; usual activities: 1=no problem, 2=moderate problems, 3= unable to do usual activities; pain and discomfort: 1=no pain or discomfort, 2=moderate pain or discomfort, 3= extreme pain or discomfort; anxiety and depression: 1=not anxious or depressed, 2=moderately anxious or depressed, 3= extremely anxious or depressed. The 5-dimensional systems are converted into a single index utility score between 0 and 1, where higher score indicated a better health state.
Time Frame: as for outcome 3
Population: FAS-DB population was analyzed. Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
units on a scale
  Change at Week 36: number analyzed (Participants) | 251 | 258
  Change at Week 36 | -0.05 (0.01) | -0.01 (0.01)
  Change at Week 48: number analyzed (Participants) | 237 | 245
  Change at Week 48 | -0.02 (0.01) | 0.00 (0.01)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline EQ-5D score as a covariate; Test type: Superiority; LS Mean Difference = -0.04, 95% CI 2-sided [-0.07 to -0.01], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline EQ-5D score as a covariate; Test type: Superiority; LS Mean Difference = -0.03, 95% CI 2-sided [-0.06 to 0.01], Standard Error of Mean 0.02

23. Secondary Outcome: Double Blind Phase: Change From Randomization in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Scores at Weeks 36 and 48
Description: The FACIT-Fatigue scale was a participant completed questionnaire consisted of 13 items that assessed fatigue. Each item was scored on a scale of 0 (maximum fatigue) to 4 (no fatigue), higher scores indicate less fatigue. Total FACIT-fatigue score was obtained by addition of scores from 13 items, giving a possible overall range from 0 (maximum fatigue) to 52 (no fatigue). Higher FACIT-fatigue scores indicated lower level of fatigue, better participant status.
Time Frame: as for outcome 3
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
units on a scale
  Change at Week 36: number analyzed (Participants) | 252 | 258
  Change at Week 36 | -0.99 (0.43) | -0.80 (0.43)
  Change at Week 48: number analyzed (Participants) | 237 | 245
  Change at Week 48 | -0.34 (0.46) | -0.52 (0.45)
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 36: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline FACIT - fatigue scale score as a covariate; Test type: Superiority; LS Mean Difference = -0.19, 95% CI 2-sided [-1.37 to 1.00], Standard Error of Mean 0.60
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Change at Week 48: Linear MMRM was used that included the fixed effects of treatment, visit, treatment-by-visit interaction, prior use of a bDMARD, and baseline FACIT - fatigue scale score as a covariate; Test type: Superiority; LS Mean Difference = 0.18, 95% CI 2-sided [-1.07 to 1.44], Standard Error of Mean 0.64

24. Secondary Outcome: Double Blind Phase: Percentage of Participants Achieving an Improvement of at Least 0.22 Units in HAQ-DI at Weeks 36 and 48
Description: HAQ-DI assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing/grooming; arising; eating; walking; reach; grip; hygiene; and other activities.. There were total of 30 items distributed in these 8 domains. Each item was scored on a 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 (least difficulty) and 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities. Percentage of participants with an improvement of at least 0.22 units in HAQ scores from baseline (Day 1) to Weeks 36 and 48 were reported in this outcome measure.
Time Frame: Baseline (Day 1), Weeks 36 and 48
Population: FAS-DB population was analyzed. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points. NRI method was used to impute missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 264 | 266
percentage of participants
  Week 36 | 67.05 | 77.07
  Week 48 | 68.56 | 75.19
Statistical Analysis 1: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 36; Test type: Superiority; Difference in percentage of participants = -10.02, 95% CI 2-sided [-17.61 to -2.42], Standard Error of Mean 3.87
Statistical Analysis 2: Comparison: Double Blind: Tofacitinib 11 mg + Methotrexate Placebo vs Double Blind: Tofacitinib 11mg + Methotrexate; Week 48; Test type: Superiority; Difference in percentage of participants = -6.62, 95% CI 2-sided [-14.26 to 1.00], Standard Error of Mean 3.89

25. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Week 52 (up to 28 days after last dose) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: For OL Phase: Baseline up to Week 24; For DB Phase: Week 24 up to Week 52 (up to 28 days after last dose)
Population: Overall study safety analysis set included all participants who received at least one dose of study drug during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label: Tofacitinib 11 mg + Methotrexate | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 694 | 264 | 266
Participants
  AEs | 362 | 107 | 109
  SAEs | 20 | 10 | 5

26. Other Pre Specified Outcome: Number of Participants With Abnormal Laboratory Parameters
Description: Abnormality criteria: Hemoglobin (Hb),Hematocrit,Erythrocytes(Ery): <0.8*LLN;Ery. Mean corpuscular volume <0.9*lower limit of normal (LLN), >1.1*upper limit of normal (ULN); Platelets:<0.5*LLN,>1.75*ULN;WBCs:<0.6*LLN,>1.5*ULN; Lymphocytes/WBCs, Neutrophils/WBCs:<0.8*LLN,>1.2* ULN;Basophils,Basophils/WBCs,Eosinophils,Eosinophils/WBCs,Monocytes, Monocytes/WBCs: >1.2*ULN;Prothrombin Time, Prothrombin Intl. Normalized Ratio:>1.1*ULN; ESR:>1.5*ULN; Bilirubin,Direct Bilirubin,Indirect Bilirubin: >1.5*ULN; Aspartate Aminotransferase (AT),Alanine AT,Gamma Glutamyl Transferase,Alkaline Phosphatase:>3.0*ULN; Protein, Albumin: <0.8*LLN, >1.2x ULN; Blood Urea Nitrogen, Creatinine, Triglycerides: >1.3*ULN;HDL Cholesterol:<0.8*LLN;Sodium <0.95*LLN, >1.05*ULN;Potassium, Chloride, Calcium, Bicarbonate: <0.9*LLN, >1.1*ULN; Glucose: <0.6*LLN, >1.5*ULN; Creatine Kinase: >2.0*ULN; Cholesterol:>1.3*ULN;Specific Gravity:<1.003;pH:<4.5; urine glucose,Ketones,urine protein,urine Hb,WBCs Esterase: >=1.
Time Frame: For OL Phase: Baseline up to Week 24; For DB Phase: Week 24 up to Week 48
Population: Overall study safety analysis Set included all participants who received at least one dose of study drug during the study. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label: Tofacitinib 11 mg + Methotrexate | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
Number analyzed (Participants) | 688 | 263 | 263
Participants | 682 | 263 | 263

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Week 52
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. AEs were evaluated for participants with at least 1 dose of the study drug during the study.
Arm/Group | Open Label: Tofacitinib 11 mg + Methotrexate | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo | Double Blind: Tofacitinib 11mg + Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/694 | 0/264 | 2/266
Serious Adverse Events (participants affected / at risk) | 20/694 | 10/264 | 5/266
Other Adverse Events (participants affected / at risk) | 158/694 | 24/264 | 31/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label: Tofacitinib 11 mg + Methotrexate (N=694) | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo (N=264) | Double Blind: Tofacitinib 11mg + Methotrexate (N=266)
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nerve root compression (Nervous system disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label: Tofacitinib 11 mg + Methotrexate (N=694) | Double Blind: Tofacitinib 11 mg + Methotrexate Placebo (N=264) | Double Blind: Tofacitinib 11mg + Methotrexate (N=266)
Bronchitis (Infections and infestations) | 0 | 3 | 7
Nasopharyngitis (Infections and infestations) | 35 | 5 | 7
Upper respiratory tract infection (Infections and infestations) | 33 | 4 | 6
Alanine aminotransferase increased (Investigations) | 16 | 5 | 10
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 16 | 0 | 0
Nausea (Gastrointestinal disorders) | 20 | 0 | 0
Headache (Nervous system disorders) | 17 | 0 | 0
Dizziness (Nervous system disorders) | 15 | 0 | 0
Hypertension (Vascular disorders) | 17 | 0 | 0
Urinary tract infection (Infections and infestations) | 19 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT02831855/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT02831855/SAP_001.pdf